CLINICAL TRIAL: NCT06936475
Title: Post-Caesarean Vaginal Cleansing With Chlorhexidine Gluconate Versus Povidone Iodine for Prevention of Endometritis: A Randomised Controlled Trial
Brief Title: Vaginal Cleansing With Chlorhexidine Versus Iodine for Prevention of Endometritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FETHA/REC/VOL2/2019/294
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Endometritis; Vaginal Cleansing; Post Caesarean
Keywords: chlorhexidine; Iodine; Endometritis; post caesarean; vaginal cleansing
MeSH Terms: conditions — Endometritis | interventions — Povidone-Iodine; Povidone; chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone group (Active Comparator): In the povidone group, vaginal cleansing was done with 3 pieces of gauze on a sponge holding forceps soaked in 30ml of 5% povidone-iodine for each patient. The soaked gauze was inserted into the vagina, rotated 360o for 30 seconds from the upper to the lower vaginal wall. This was done when clots had been evacuated from the vagina with dry gauze on a sponge holding forceps according to departmental protocol.
  Interventions: Drug: Povidone-Iodine
- Chlorhexidine group (Experimental): In the chlorhexidine group, vaginal cleansing was done with 3 pieces of gauze on a sponge holding forceps soaked in 30ml of 0.5% chlorhexidine for each patient. The soaked gauze was inserted into the vagina, rotated 360o for 30 seconds from the upper to the lower vaginal wall. This was done when clots had been evacuated from the vagina with dry gauze on a sponge holding forceps according to departmental protocol.
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Povidone-Iodine — 5% povidone iodine
  Other Names: Povidone
  Arms: Povidone group
Drug: Chlorhexidine Gluconate — 0.5% chlorhexidine
  Other Names: Chlorhexidine
  Arms: Chlorhexidine group

SUMMARY:
Povidone has been approved for vaginal cleansing in the prevention of endometritis postcaesarean section. chlorhexidine solution which is cheap and readily available as shown to prevent endometritis.The aim of this study is to compare the effectiveness of post-operative vaginal cleansing with povidone-iodine versus chlorhexidinegluconate in reducing post-caesarean maternal endometritis

DETAILED DESCRIPTION:
BACKGROUND: Maternal infectious morbidity is a common complication of caesarean section and is the third leading cause of maternal mortality in Nigeria. It accounts for 15% of maternal death worldwide. Post-caesarean maternal infectious morbidity (endometritis) is still a big challenge despite prophylactic antibiotics and other modalities adopted to prevent it. Recently, preoperative vaginal cleansing with povidone-iodine was conditionally recommended in reduction of post-caesarean endometritis by WHO but in some emergent conditions, the practice may not be feasible. There is need to research effective post-caesarean vaginal cleansing antiseptic agents which may offer benefits in such emergent conditions.

AIM: To compare the effectiveness of post-operative vaginal cleansing with povidone-iodine versus chlorhexidinegluconate in reducing post-caesarean maternal endometritis at the Alex Ekwueme Federal University Teaching Hospital Abakaliki (AEFUTHA).

METHODOLOGY: This was a single blinded randomized controlled trial involving two hundred and forty four (244) consenting pregnant women booked for emergency lower segment Caesarean section at AEFUTHA and Mile 4 Hospital, Abakaliki; with 122 women randomized into the Povidone-iodine arm (control arm) and 122 into the Chlorhexidinegluconate arm. Both groups received prophylactic antibiotics and anterior abdominal wall scrubbing. The control group received post-operative vaginal cleansing with Povidone iodine while study group received chlorhexidinegluconate. immediately after skin closure. Subsequently, they were reviewed for endometritis daily till discharge or up to 7 days for patients who had the need to stay up to 7 days or beyond. Data was analyzed using statistical Package for Social Science (IBM SPSS) software (version 24, Chicago II, USA). Continuous variables were presented as mean and standard deviation (Mean ± 2SD), while categorical variables were presented as numbers, frequencies and percentages. Student t test was used for comparison between groups for continuous variables and mean of the two groups. Chi-square test was used for comparison between groups for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women at > 28 weeks gestational age undergoing emergency caesarean section.
* Emergency caesarean sections for women in labour, with ruptured membrane or cord prolapse.
* Pregnant women that gave consent to participate in the study

Exclusion Criteria:

* Elective caesarean sections
* Known allergy to povidone iodine or chlorhexidinegluconate
* Diabetes mellitus/ glucose intolerance undergoing elective caesarean section.
* Asymptomatic placenta praevia undergoing elective caesarean section
* Patients who have chorioamnionitis
* Immunosuppressive conditions like AIDS, steroid use
* Patients who have coexisting uterine fibroid.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 239 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
post caesarean endometritis | 7 days
  the number of participants that will develop endometritis following use of either agents

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No
This will be made available following publication